CLINICAL TRIAL: NCT06730256
Title: A Clinical Study to Explore the Safety, Efficacy, and Pharmacokinetics of CT0596 CAR-T Cell Injection in Patients With Relapsed/Refractory Multiple Myeloma and Relapsed/Refractory Plasma Cell Leukemia
Brief Title: A Study of CT0596 in Relapsed/Refractory Multiple Myeloma and Relapsed/ Refractory Plasma Cell Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT0596-CG6022_02
Record Dates: First submitted 2024-12-04; First posted 2024-12-12 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory Plasma Cell Leukemia; Relapsed/Refractory Multiple Myeloma
Keywords: Relapsed/Refractory Multiple Myeloma; Relapsed or Refractory Plasma Cell Leukemia; CAR-T
MeSH Terms: conditions — Leukemia, Plasma Cell; Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T cells Infusion chimeric antigen receptor T cells (Experimental): Drug: CAR-T cells Infusion chimeric antigen receptor T cells
  Interventions: Drug: CAR-T cells Infusion chimeric antigen receptor T cells

INTERVENTIONS:
Drug: CAR-T cells Infusion chimeric antigen receptor T cells — CAR-T cells Infusion chimeric antigen receptor T cells

SUMMARY:
A Clinical Study to Explore the Safety, Efficacy, and Cellular Metabolic Dynamics of CT0596 CAR-T Cell Injection in Patients With Relapsed/Refractory Multiple Myeloma and Plasma Cell Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria to be enrolled:

  1. Patients must voluntarily sign the informed consent form (ICF) and must be willing and be able to adhere to the trial visit schedule and other protocol requirements and agree to be in long term follow-up (LTFU) for up to 15 years as mandated by the regulatory guidelines.
  2. Age ≥ 18 years;
  3. Patients with R/RMM who have received at least 3 prior lines of therapy, including at least 1 proteasome inhibitor and at least 1 immunomodulator (IMiD). Patients with RRpPCL had received at least 1 prior line of therapy. Number of lines of therapy was defined according to the guidelines provided in Rajkuma[1]r 2015 . Patients must have received at least 1 complete cycle of therapy for each line of therapy.
  4. According to multiple myeloma IMWG 2016 and plasma cell leukemia IMWG 2013, patients must have progressive disease following or during the last treatment.
  5. Patients must have measurable disease based on at least one of the following parameters:
  6. Expected survival > 12 weeks;
  7. Eastern Cooperative Oncology Group (ECOG) score 0- 1 ;
  8. Patients should meet the following test results
  9. Female patients of childbearing potential must have a negative pregnancy test at screening and prior to receiving lymphodepletion therapy and are willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment and are absolutely prohibited from donating eggs for 1 year after receiving study treatment infusion during the study ;Male patients are willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment if they are sexually active with a female of childbearing potential. Sperm donation is absolutely prohibited within 1 year following study treatment infusion for all male patients during the study.

Exclusion Criteria:

* 1. Pregnant or lactating women; 2. Patient has any significant condition(s), laboratory abnormality or psychiatric illness that would impair the ability of the patient to receive or tolerate the planned treatment or in the opinion of the investigator, participation would not be in the best interest of the patient (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments 3. Patients seropositive for HIV, active hepatitis C virus (HCV), or active hepatitis B virus (HBV) infection. History of treated hepatitis B or C is permitted if the viral load is undetectable per qPCR and or nucleic acid testing; 4. Patients with any uncontrolled active infection, including but not limited to patients with active tuberculosis (investigator 's judgment); 5. Toxicities caused by previous treatment have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) ≤ Grade 1, except alopecia and other events that are judged tolerable by the investigator; 6. Previous allogeneic stem cell transplantation; autologous stem cell transplantation within 12 weeks prior to signing informed consent; 7. Have received treatment for the disease within 14 days before informed consent 8. Have received cell therapy within 28 days before informed consent. 9. Systemic glucocorticoids equivalent to > 15 mg/day prednisone within 7 days prior to informed consent, with the exception of topical glucocorticoids; 10. Vaccination with live attenuated vaccines , inactivated vaccines or RNA vaccines within 4 weeks prior to informed consent; 11. Allergic or intolerant to lymphodepletion, tocilizumab, or allergic to components (DMSO) in CT0596 CART cell infusion preparation; or previous history of other serious allergies such as anaphylactic shock; 12. Patients with secondary plasma cell leukemia, Waldenström macroglobulinemia, POEMS syndrome, or primary light chain amyloidosis at Screening; 13. Patients with any of the following cardiac conditions within 6 months prior to screening: 14. Patients who require supplemental oxygen to maintain oxygen saturation > 92%; or Patients with known or suspected COPD who have Forced Expiratory Volume in 1 second (FEV1) < 50% of predicted normal on spirometry; 15. Patients with active autoimmune diseases, including but not limited to psoriasis, rheumatoid arthritis and other diseases requiring long-term immunosuppressive therapy; 16. Patients with second primary malignancies in addition to MM are not eligible if the second primary malignancy has required treatment within the past 2 years or is not in complete remission. Exceptions include the following that have been successfully treated - nonmetastatic basal cell or squamous cell skin carcinoma, non-metastatic prostate cancer, carcinoma-in-situ of breast or cervix, non-muscle invasive bladder cancer 17. Patients with symptomatic central nervous system (CNS) disease or suspected CNS metastases; 18. Major surgery within 2 weeks before informed consent or planned during the study period or within 4 weeks after giving study treatment (excluding local anesthesia such as cataract)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2027-01-03 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) after CT0596 infusion | 12 months after CT0596 infusion]
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria
Maximum tolerated dose and/or dose range | 12 months after CT0596 infusion
  Evaluate Dose limited toxicity and recommended dosage range after CT0596 infusion

SECONDARY OUTCOMES:
Overall response rate (ORR) as assessed by the investigator | 12 months after CT0596 infusion
  Overall response rate (ORR) defined as proportion of patients achieving partial response or better based on International Myeloma Working Group defined response criteria
Complete response/stringent complete response (CR/sCR) rate | 12 months after CT0596 infusion
  Rate of complete response/stringent complete response (CR/sCR) defined as proportion of patients achieving complete response or better based on International Myeloma Working Group（ IMWG） defined response criteria.
Rate of very good partial response (VGPR) and above | 12 months after CT0596 infusion
  Rate of complete very good partial response response/stringent complete response (VGPR/CR/sCR) defined as proportion of patients achieving VGPR or better based on International Myeloma Working Group（IMWG） defined response criteria
Duration of response (DOR) | 12 months after CT0596 infusion
  Duration of response （DOR） is defined as the time from first achievingpartial response（ PR ）or better to confirmed disease progression or death from any cause
Minimal residual disease (MRD) negative rate | 12 months after CT0596 infusion
  Minimal residual disease (MRD) negative rate is defined as the proportion of patients with VGPR or better who achieved 10-5 sensitivity of nucleated cell
Time to response (TTR) | 12 months after CT0596 infusion
  Time to response（TTR ）defined as the time from the date of apheresis to the date of initial assessment of PR or better according to IMWG2016 criteria
Progression-free survival (PFS) | 12 months after CT0596 infusion
  Progression-free survival（PFS） defined as the time from the date of apheresis of the subject to the first assessment of confirmed disease progression or death from any cause according to International Myeloma Working Group（ IMWG）2016 criteria, whichever occurs first.
Test Copy number of CAR | 12 months after CT0596 infusion]
  Evaluate cellular pharmacokinetics of CT0596
Overall survival (OS) | 12 months after CT0596 infusion
  Overall survival（OS） defined as the time from the date of apheresis of the subject to death from any cause
Cytokines in the peripheral blood after CT0596 infusion | 12 months after CT0596 infusion]
  Serum concentrations of interleukin (IL)-6 after CT0596 infusion

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No